CLINICAL TRIAL: NCT05803304
Title: Efficacy of a Novel Web-based Physical Activity Intervention Designed to Promote Adherence to Physical Activity Guidelines in Adults With Obesity
Brief Title: Web-based Physical Activity Intervention to Promote Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacob Kariuki, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00005168; 7R56HL164737-02 (NIH)
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
Keywords: Physical activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Intervention (Experimental): Insufficiently active adults with obesity assigned to the PATH intervention.
  Interventions: Behavioral: PATH Intervention; Other: Physical activity tracker; Behavioral: Dietary education
- Attention Control Group (Active Comparator): Insufficiently active adults with obesity assigned to the attention control group. At the end of the 6-month study period, participants will receive access to the PATH program, without the coaching component.
  Interventions: Behavioral: Attention Control Intervention; Other: Physical activity tracker; Behavioral: Dietary education

INTERVENTIONS:
Behavioral: PATH Intervention — The PATH intervention guides participants in making changes in their lifestyle and PA habits to support long-term adherence to the minimum threshold of PA Guidelines (150 MVPA minutes per week). The health coach provides participants with access the PATH website and a detailed orientation on how to use the resources included in PATH. The health coach meets remotely with each participant twice per month to develop a tailored plan geared towards increasing MVPA by about 10 minutes per week. The PA prescription process begins by identifying a suitable PATH level for each participant. After assigning the PATH level, the health coach guides each participant in selecting their weekly PA goal and helps them start slowly with a plan to establish regular exercise frequencies of 3-5 days per week. The coach also guides participants to select activities with intensity to help them progress along the PA continuum (i.e., from inactive to light PA and then MVPA).
  Arms: PATH Intervention
Behavioral: Attention Control Intervention — A health coach will have a zoom meeting with each control group participant where they will be provided with an electronic copy of the "Be Active Your Way" booklet, developed by the Centers for Disease Control and Prevention (CDC) to help individuals integrate PA into their daily lives. The coach will orient the participant to the key strategies used in the booklet and encouraged them to use it regularly and to self-monitor PA using the Fitbit during the entire course of the study. In addition, the group will be introduced to www.health.com, a jargon free website that focuses on general health topics and latest medical news. At the end of the meeting, the participants will be asked to provide a schedule for zoom meetings the study team twice per month during the 6 month study. The meetings will focus on their progress in using the "Be Active Your Way" handout and the health.com website.
  Arms: Attention Control Group
Other: Physical activity tracker — Participants will be asked to wear Fitbit Charge 5 on their non-dominant hand for the entire duration of the study using a 24hr wear protocol.
  Other Names: Fitbit
Behavioral: Dietary education — Diet quality and barriers to healthy eating will be evaluated at baseline, and then all study participants will be provided with educational materials that are curated to promote diet quality. Participants will receive a monthly email with a brief PDF addressing a diet component focused on improving diet quality to reduce CVD risk and improve general health.

SUMMARY:
In this study insufficiently active adults with obesity will be assigned to either the Physical Activity for The Heart (PATH) intervention or an attention control group.

DETAILED DESCRIPTION:
The United States' 2018 Physical Activity Guidelines recommend that American adults should achieve ≥150 min of moderate intensity physical activity (PA), 75 min of vigorous PA, or an equivalent combination of both moderate and vigorous physical activity (MVPA) weekly. Yet, adherence to these Guidelines is low, with 26% of adults with normal weight and 14% of adults with obesity attaining the minimum recommended PA levels. The low PA levels are associated with the rising prevalence of obesity and increase the relative risk of stroke, coronary heart disease, and diabetes by 60%2, 45%, and 30%, respectively. Since individuals with obesity are more vulnerable to cardiovascular disease (CVD) and its risk factors, weight loss is recommended. Yet, even without weight-loss, PA significantly reduces CVD risk. However, individuals with obesity face complex multifaceted barriers that reduce their engagement in PA.

Barriers to PA associated with obesity include stigma, shame, poor fitness, and low self-efficacy. These evoke fear of embarrassment and pain, contributing to aversion of PA. To mitigate these barriers, web-based PA programs targeting adults with obesity have been developed. Preliminary data suggest improved retention, but the effects on PA are heterogeneous. Limitations of these interventions include lack of human contact, 'one-size-fits-all' strategies, unmet weight-loss expectations, and generic content that fails to address the barriers associated with obesity. Researchers have reported that individuals with obesity prefer programs that are convenient, fun to engage in, and feature people who they can relate to in body size, fitness level, and age. Yet, there is a paucity of PA interventions intentionally designed to flexibly incorporate these preferences.

To address the limitations of previous interventions, the research team of this study designed the web-based Physical Activity for The Heart (PATH) intervention. PATH leverages openly accessible platforms, such as YouTube, to provide workout videos that match the specific preferences expressed in our formative studies and the extant literature. In developing PATH, the researchers employed an iterative bottom-up approach where the target population was engaged in the selection and rating of the workout videos. Then, highly rated workouts (≥3.5/5 stars) were vetted by the study team for content relevance and safety, and then curated on the PATH website in 3 intensity levels (beginner, intermediate, proficient) to foster gradual progression from low to high intensity PA. The researchers added backend features that enable a remote health coach to help users set their PA goals and select a PA regimen that is safe for their fitness level. Each PATH user has a personalized dashboard displaying their recommended workouts and progress towards their PA goals.

In this study, 88 insufficiently active adults with obesity will be assigned to either the PATH intervention or the attention control group for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Regular access to the Internet
* BMI ≥30kg/m^2
* Successful self-monitoring of PA (≥4 days with ≥10hrs wear time) via waist worn Actigraph
* Non-adherence to the PA Guidelines (<150 min of MVPA/wk)

Exclusion Criteria:

* Pregnancy or intention to become pregnant within 6 months
* Mobility restrictions, or any condition that requires supervised PA (e.g., stroke)
* Individuals with history of heart disease, diabetes, or those who respond in affirmative to any question in the Physical Activity Readiness Questionnaire will be required to obtain Primary Care Provider (PCP) clearance before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Weekly Moderate-to-Vigorous Physical Activity | Baseline, Month 6
  Participants will wear a physical activity tracker around their waist for 7 days to assess the number of minutes of MVPA.
Change in Number of Participants Adhering to PA Guidelines | Baseline, Month 6
  Adherence to PA Guidelines will be defined as achieving ≥150 min of MVPA per week. Percent change in adherence is calculated as: [(Post-intervention MVPA - Baseline MVPA)/Recommended MVPA×100].
Change in Step Count | Baseline, Month 6
  Daily step count will be measured with a physical activity tracker worn on the wrist for at least 10 hours per day while awake.
Change in 2013 Atherosclerotic Cardiovascular Disease (ASCVD) Risk Calculator | Baseline, Month 6
  The algorithm provides sex and race-specific estimates for the first CVD event for black and white men and women. The scores range from 0-100% with higher scores representing poor cardiovascular health status. The between group difference in risk score change is computed as the end of study score minus the baseline score.

SECONDARY OUTCOMES:
Change in Waist Circumference | Baseline, Month 6
  Waist circumference is measured in centimeters (cm).
Change in Weight | Baseline, Month 6
  Weight is measured in kilograms (kg).
Change in Systolic Blood Pressure | Baseline, Month 6
  Systolic blood pressure is the amount of pressure the heart generates when pumping blood through the arteries to the body. Normal systolic blood pressure as lower than 120 millimeters of mercury (mmHg).
Change in Diastolic Blood Pressure | Baseline, Month 6
  Diastolic blood pressure is the amount of pressure in your arteries when your heart is at rest between beats. Normal diastolic blood pressure as lower than 80 mmHg.
Change in Life's Essential 8™ Score | Baseline, Month 6
  Life's Essential 8 is a way to assess cardiovascular health developed by the American Heart Association. Life's Essential 8 has 8 components: diet, physical activity, exposure to nicotine, sleep, body mass index (BMI), blood lipids, blood glucose, and blood pressure. Each component is scored with an algorithm and scores range from 0 to 100. A composite score of overall cardiovascular health can be generated and it also ranges from 0 to 100. A score of 0 indicates a low health score, a score of 50 indicates moderate health, and a score of 100 is the highest health for each of the 8 components as well as the overall score.
Change in Hemoglobin A1c | Baseline, Month 6
  The hemoglobin A1c test result reflects average blood sugar level over the past three months. Specifically, the A1c test measures what percentage of hemoglobin is coated with sugar (glycated). Values below 5.7% are normal, values between 5.7% and 6.4% indicate prediabetes, and values of 6.5% and higher indicate diabetes.
Change in Adiponectin | Baseline, Month 6
  Adiponectin is a hormone released by adipose tissue, and other body tissues, that assists with insulin sensitivity and reducing inflammation. Normal ranges vary depending on sex and BMI and in general lower levels are associated with health conditions of obesity, Type 2 diabetes, and atherosclerosis. In people with a BMI of less than 25, the normal range for males and females is 5 to 37 micrograms per milliliter (µg/mL). In those with a BMI of 25 to 30 the normal range for males is 5 to 28 µg/mL and the normal range for females is 4 to 20 µg/mL. In people with a BMI over 30 the normal range for males is 2 to 20 µg/mL and the normal range for females is 4 to 22 µg/mL.
Change in Total Cholesterol | Baseline, Month 6
  Cholesterol is waxy substance which is produced by the liver or comes from food that is consumed. Cholesterol concentrations are commonly used as a marker for cardiovascular disease risk. Healthy levels of total cholesterol are 125 to 200 milligrams (mg) per deciliter (dL).
Change in Low-density Lipoprotein (LDL) Cholesterol | Baseline, Month 6
  Healthy levels of LDL cholesterol are below 100mg/dL.
Change in High-density Lipoprotein (HDL) Cholesterol | Baseline, Month 6
  HDL cholesterol is the "good" cholesterol because it is a type of fat that removes cholesterol from blood, thereby preventing build up. Healthy levels for HDL cholesterol are 40mg/dL or higher in adult males and 50 mg/dL or higher in adult females.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kariuki, PhD, NP, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available for the main study outcomes. Other data from the questionnaires or other assessments may be available for sharing on a case by case basis.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing one year after publication of study outcomes.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposal should be directed to jacob.kariuki@emory.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Derived] Kariuki J, Burke L, Erickson K, Sereika S, Paul S, Cheng J, Biza H, Abdirahman A, Wilbraham K, Milton H, Brown C, Sells M, Osei Baah F, Wells J, Chandler R, Barone Gibbs B. Acceptability and Preliminary Efficacy of a Novel Web-Based Physical Activity for the Heart (PATH) Intervention Designed to Promote Physical Activity in Adults With Obesity: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 18;14:e67972. doi: 10.2196/67972. PMID 40101744

DOCUMENTS (1):
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT05803304/ICF_000.pdf